CLINICAL TRIAL: NCT05474885
Title: BCMA-CD19 cCAR T Cell Treatment of Relapsed/Refractory Systemic Lupus Erythematosus (SLE)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCAR Bio Therapeutics Ltd. China (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG180-001
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-04

CONDITIONS: Relapsed/Refractory, Systemic Lupus Erythematosus (SLE)
Keywords: BCMA-CA19 CAR; lupus; SLE; systemic lupus erythematosus; autoimmune disorders
MeSH Terms: conditions — Recurrence; Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA-CD19 cCAR T cells (Experimental): Dose escalation phase: patient's T cells will be transduced with a lentiviral vector to express a BCMA-CD19 cCAR. with an escalation approach.
  Interventions: Biological: BCMA-CD19 cCAR T cells

INTERVENTIONS:
Biological: BCMA-CD19 cCAR T cells — BCMA-CD19 cCAR T cells are used to treat patients. Patient will be administered either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of BCMA-CD19 cCAR T cells in patients with relapsed and/or refractory SLE.

DETAILED DESCRIPTION:
Systemic lupus erythematous (SLE) is a chronic diffuse connective tissue disease with unexplained etiology that can involve multiple systems in the body. SLE is considered as an incurable disease and traditional SLE treatment aims at long-term remission. Glucocorticoids combined with immunosuppressive agents are still the main treatment strategies. Recently, biological agents targeting abnormal immune cells, such as rituximab and belimumab, which deplete B cells have also achieved some success in the treatment of SLE. However, these agents cannot permanently reverse the production of abnormal antibodies as they are unable to eliminate pathogenic long-lived plasma cells. The BCMA-CD19 CAR T-cells are designed to deplete antibody-producing 'root", B cells and plasma cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~65 years old;
2. Expected survival period ≥ 3 months;
3. Serum creatinine <221.0μmol/L (2.5mg/dl);
4. AST/ALT below 3 times the upper limit of normal, blood bilirubin <34.2 μmol/L (2.0 mg/dl);
5. Cardiopulmonary function is basically normal, echocardiography indicates that the ejection fraction is >50%, and the oxygen saturation is above 94% in the resting state without oxygen;
6. No obvious active infection;
7. Physical fitness score 0~2 points (ECOG standard);
8. There are suitable veins for blood cell apheresis or whole blood collection, and there are no contraindications for blood collection;
9. Since the effect of CAR T cell therapy on the fetus is unknown, women of childbearing age should have a negative serum or urine pregnancy test 48 hours before CAR T cell reinfusion, and agree to take effective measures during the trial until the last follow-up. contraceptive measures;
10. Voluntary participation and informed consent signed by the patient or his/her legal/authorized representative.

Exclusion Criteria:

1. Severe systemic lupus erythematosus: BILAG score at least 1 system is A and (or) >2 systems reach B, or SELENA SLEDAI>12 points.
2. CNS disease: Active central nervous system (CNS) lupus (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident [CVA], encephalitis or CNS vasculitis), visual Disorders, cranial neuropathy requiring intervention
3. Abnormal liver function: aspartate transaminase (AST) or alanine transaminase (ALT) or glutamyl transpeptidase (GGT) detection value is greater than 3 times the upper limit of normal (ULN); or alkaline phosphatase ( ALP) or total bilirubin test value greater than 1.5 times the upper limit of normal (ULN);
4. Kidney disease: hemodialysis or high-dose glucocorticoid treatment is required within 90 days before visit 2, such as prednisone (or equivalent dose of glucocorticoid) ≥ 100 mg/d, or creatinine (Cr) or blood urea nitrogen (BUN) detection value greater than 1.5 times the upper limit of normal (ULN), or eGFR ≤ 60ml/min before visit 2. eGFR is calculated using the MDRD formula: eGFR (ml/min×1.73m^2)=186×serum creatinine (Scr)-1.154×age-0.203× (multiply by 0.724 if the subject is a female)
5. Cardiovascular disease: history of acute myocardial infarction, or unstable angina pectoris, severe arrhythmia (multi-source frequent premature ventricular tachycardia, ventricular tachycardia, ventricular fibrillation) in the past 6 months; New York heart function class (NYHA) class III- Level IV
6. Other uncontrolled diseases: acute or chronic diseases (such as acute pneumonia, pulmonary hypertension, diabetic ketoacidosis, acute pancreatitis, etc.) that are clinically unstable or have not been effectively controlled and are not related to SLE. judgments that may confound study results or place subjects at undue risk.
7. Infection: Subject has acute or chronic infection requiring treatment (eg, tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria)
8. Surgery or other conditions: planning to undergo surgery or have any other medical history (eg, recent history of sepsis), abnormal laboratory tests, or other conditions, judged by the investigator to be inappropriate to participate in this study
9. Biologics therapy: Received any drug therapy (antibody, inhibitor or agonist) targeting T, B lymphocytes, cytokines or receptors within two months
10. Participated in any clinical study within 3 months prior to enrollment
11. The use of contraindicated drugs or therapies may affect the judgment of the efficacy of CART: 1) Received any of the following treatments within 90 days before Visit 2: (1) Intravenous immune globulin (IVIG); (2) Oral high-dose glucocorticoids Hormones, such as prednisone >100mg/d; (3) plasma exchange, leukotomy; 2) new immunosuppressive/immune modulators were added within 60 days before visit 2, and the disease is still under control.
12. Received live vaccine treatment within 30 days prior to Visit 2
13. Transplantation: History of vital organ transplantation (eg, heart, lung, kidney, liver) or hematopoietic stem cell/or bone marrow transplantation
14. HIV positive.
15. Active hepatitis B or C.
16. Suffering from malignant tumors of other organs at the same time.
17. Pregnant or lactating women.
18. Inability to understand or follow the research protocol.
19. Participate in other clinical investigators during the same period.
20. Have any other clinically significant disease history or current disease that, in the judgment of the research physician, may pose a risk to the safety of the subjects, or interfere with the completion of the research procedure and the evaluation of safety and efficacy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The number and incidence of adverse events after BCMA-CD19 cCAR T cell infusion | 3 months after CAR infusion
  Evaluation all possible adverse reactions, including the number, incidence, and severity of symptoms such as cytokine release syndromes and neurotoxicity within 3 months after CAR infusion.

SECONDARY OUTCOMES:
Autoantibody detection | 6 months after CAR infusion
  Autoantibody detection up to 6 months after BCMA-CD19 cCAR T cells infusion
SLEAI score | 2 years after CAR infusion
  SLEAI score taken up to 2 years after BCMA-CD19 cCAR T cells infusion
Renal functions | 1 year after CAR infusion
  Renal functions monitored up to 1years after BCMA-CD19 cCAR T cells infusion
Disease control | 2 years after CAR infusion
  Disease control monitored up to 2 years after BCMA-CD19 cCAR T cells infusion)
Overall survival | 2 years after CAR infusion
  Overall survival (2 year after CAR infusion). The time from the start of BCMA-CD19 cCAR infusion to death is determined as the overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan People's Hospital, Zhongshan, Guangdong, China